CLINICAL TRIAL: NCT05353582
Title: Preoperative Systemic Therapy With FOLFOXIRI Plus Bevacizumab Followed by Cytoreductive Surgery Versus Upfront Cytoreductive Surgery for Resectable Colorectal Peritoneal Metastases: A Randomized Phase 2 Trial
Brief Title: Preoperative Systemic Therapy for Colorectal Cancer Peritoneal Metastases
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanhong Deng, Director, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUCS
Record Dates: First submitted 2022-04-22; First posted 2022-04-29 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Colorectal Neoplasms; Colorectal Cancer; Colorectal Cancer Metastatic; Peritoneal Metastases; Peritoneal Cancer; Peritoneal Neoplasms; Chemotherapy Effect; Cytoreductive Surgery; Hyperthermic Intraperitoneal Chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy group (Experimental): 6 cycles of mFOLFOXIRI±Bev is followed by cytoreductive surgery. Postoperative 6 cycles of mFOLFOX is scheduled.
  Interventions: Drug: Preoperative systematic therapy; Procedure: CRS+HIPEC; Drug: Postoperative chemotherapy
- Upfront surgery group (Active Comparator): Upfront surgery group is followed by 12 cycles of mFOLFOX+Bev
  Interventions: Procedure: CRS+HIPEC; Drug: Postoperative chemotherapy

INTERVENTIONS:
Drug: Preoperative systematic therapy — 6 cycles of mFOLFOXIRI±Bev is administrated before CRS+HIPEC. Irinotecan165mg/m2 IV day 1, oxaliplatin 85mg/m2 IV day 1, leucovorin 400mg/m2 IV day , bevacizumab mg/kg IV day 1, 5-fluorouracil 400mg/m2, continuous infusion over 46-48h. Dose reduction is permitted. Bev will not be administrated in at the last two cycles for minimizing surgery complications.
  Arms: Chemotherapy group
Procedure: CRS+HIPEC — CRS+HIPEC aims to achieve CC0/CC1 resection. Oxaliplatin or mitomycin C is determined by the treating physician.
Drug: Postoperative chemotherapy — 6 cycles of mFOLFOX+Bev is administrated after CRS+HIPEC. Oxaliplatin 85mg/m2 IV day 1, leucovorin 400mg/m2 IV day , bevacizumab mg/kg IV day 1, 5-fluorouracil 400mg/m2 IV bolus day 1,5-fluorouracil 400mg/m2, continuous infusion over 46-48h. Dose reduction is permitted.
  Arms: Chemotherapy group
Drug: Postoperative chemotherapy — 12 cycles of mFOLFOX+Bev is administrated after CRS+HIPEC. Oxaliplatin 85mg/m2 IV day 1, leucovorin 400mg/m2 IV day , bevacizumab mg/kg IV day 1, 5-fluorouracil 400mg/m2 IV bolus day 1,5-fluorouracil 400mg/m2, continuous infusion over 46-48h. Dose reduction is permitted.
  Arms: Upfront surgery group

SUMMARY:
This is an open-label, parallel-group, phase 2 randomized trial which randomizes patients with isolated resectable colorectal cancer peritoneal metastases to receive preoperative systematic therapy followed by CRS+HIPEC and postoperative chemotherapy or upfront CRS+HIPEC followed by postoperative chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1;
* Historically and radiologically confirmed colorectal cancer peritoneal metastasis except for appendical origin;
* Tolerable to scheduled chemotherapy;
* No evidence of extraperitoneal metastases at enrollment;
* Resectable disease determined by radiological and laparoscopy/laparotomy;
* No systematic therapy within 6 months before enrollment;
* Tolerable to cytoreductive surgery.

Exclusion Criteria:

* Without adequate organ function (e.g. :neutrophil countt≤1.5×10^9/L, or platelets≤75×10^12/L，or hemoglobin<90g/L, or aminotransferase、aspartate aminotransferaseAST<2.5ULN, or total bilirubin<1.5ULN, or creatinine<1.5ULN;
* Emergency surgery;
* Recent thromboembolic event or cerebrovascular disease (12 months before enrollment);
* Pregnancy or lactation
* Comorbid with severe physical or mental disease.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-06-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | Up to five years after randomization
  From randomization to progression by RECIST1.1, or appearance of measurable lesion after non-measureable lesion, or intraoperative unresectable disease, or recurrence after surgery, or death from any reason.

SECONDARY OUTCOMES:
Response to preoperative systematic therapy | About 4 months after randomization
  Assessed by tumor regression grade
Major adverse events of systematic therapy | Up to 8 months after randomization
  Grade ≥3 adverse events by CTCAE 5.0
Overall survival | Up to five years after randomization
  From randomization to death of any cause
Intraoperative peritoneal cancer index | About 4 months after randomization
  Peritoneal cancer index (PCI) is a tool which sum scores in thirteen abdominal regions according to tumor size.
Complete cytoreductive surgery | About 4 months after randomization
  R0/R1 resection or CC0/CC1 resection
Hospitalization time | About 4 months after randomization
  Safety of cytoreductive surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Participant-level raw data will not publically available unless reasonable request.